CLINICAL TRIAL: NCT02267057
Title: Efficacy of Pain Treatment on Depression in Patients With Dementia. A Randomized Clinical Trial.
Brief Title: Efficacy of Pain Treatment on Depression in Patients With Dementia
Acronym: DEP-PAIN-DEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Bettina Husebo, MD, assoc prof. University of Bergen, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFR project nr 221951; 2013-002226-23 (EudraCT Number)
Record Dates: First submitted 2014-07-07; First posted 2014-10-17 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Depression; Pain; Dementia
Keywords: Pain measurement; Pain assessment; Pain management; Analgesia; Analgesics; Depressive symptoms; Alzheimer disease; Vascular dementia; Multi-infarct dementia; Frontotemporal lobar degeneration; Lewy body disease
MeSH Terms: conditions — Depression; Pain; Dementia; Agnosia; Alzheimer Disease; Dementia, Vascular; Dementia, Multi-Infarct; Frontotemporal Lobar Degeneration; Lewy Body Disease | interventions — Acetaminophen; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol or buprenorphine treatment (Active Comparator): Paracetamol tablets 1 g three times daily or Buprenorphine transdermal system 5 micrograms/hour every 7 days, may be titrated up to 10 micrograms/hour every 7 days if clinically appropriate.
  Interventions: Drug: Paracetamol; Drug: Buprenorphine
- Paracetamol placebo or buprenorphine placebo (Placebo Comparator): Paracetamol placebo tablet three times daily or buprenorphine transdermal system placebo every 7 days.
  Interventions: Drug: Paracetamol placebo; Drug: Buprenorphine placebo

INTERVENTIONS:
Drug: Paracetamol — Paracetamol granulate supplied by Weifa (Paracet) and 1 g paracetamol tablets produced by Kragerø tablettproduksjon for blinding purposes.
  Other Names: Paracet (Weifa)
  Arms: Paracetamol or buprenorphine treatment
Drug: Buprenorphine — Buprenorphine 5 micrograms/hour and 10 micrograms/hour transdermal system produced by Mundipharma, identical to placebo transdermal system.
  Other Names: Norspan (Mundipharma)
  Arms: Paracetamol or buprenorphine treatment
Drug: Paracetamol placebo — Paracetamol placebo tablets produced by Kragerø tablettproduksjon.
  Arms: Paracetamol placebo or buprenorphine placebo
Drug: Buprenorphine placebo — Buprenorphine transdermal system placebo produced by Mundipharma.
  Arms: Paracetamol placebo or buprenorphine placebo

SUMMARY:
The purpose of this study is to determine whether pain treatment can reduce symptoms of depression in patients suffering from dementia and depression. Depression is commonly diagnosed in patients with dementia. If the investigators find a reduction in depressive symptoms when pain treatment is applied, this will support the hypothesis that undiagnosed pain may present itself as depression in patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in long term nursing home units for at least 4 weeks prior to study
* Diagnosed with probable or possible dementia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), FAST score > 4
* Diagnosed with depression ≥ 4 week duration as measured by CSDD ≥ 8
* Written, informed consent provided by the participant (if they have capacity) or assent (if they do not have capacity) and a written proxy informed consent from a legally authorized representative empowered to make health-related decisions for the potential study participant

Exclusion Criteria:

* The patient is contra-indicated to study drugs of pain treatment, in another trial, or had no carer.
* Participants are ineligible if they are clinical critical (e.g. suicide risk)
* Clinician responsible for care, or study clinician considers that the patient suffers from any physical condition, which would make participation in the trial distressing or likely to increase suffering
* Advanced severe medical disease/disorder with expected survival less than 6 months or that could interfere with participation
* Psychosis or other severe mental disorder prior to dementia diagnosis
* Severe aggression (≥8) on item 3 of the NPI subscale, with aggression as the predominant symptom
* Schizophrenia, schizoaffective disorder and bipolar disorder
* Uncontrolled epilepsy
* Severe liver impairment
* Renal failure
* Severe injury or anaemia (Hb < 8.5 mmol/l), comatose state, current enrolment in another experimental protocol
* Known allergy or adverse reaction to paracetamol or buprenorphine transdermal patch
* Advanced severe medical disease with expected survival of less than six months, severe psychiatric or neurological disorder.
* Patients with diseases that make it impossible to follow the research schedule are excluded

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-08; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Change in the Cornell Scale for Depression in Dementia (CSDD) | Week -2, week 0, week 6 and week 13

SECONDARY OUTCOMES:
Change in actigraphy recorded sleep patterns and circadian rhythm | Week -1 to 0 and week 12 to 13
  Actigraph will be used for a period of 1 week before study treatment starts, and in the last week of treatment, on a selection of patients in the placebo group and in the treatment group.
Change in the Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) | Week -1, week 0, week 6 and week 13
Change in the Mini-Mental State Examination (MMSE) | Week -1 and week 13
Change in the Mobilization- Observation - Behavior - Intensity - Dementia-2 (MOBID-2) Pain Scale | Week -1, week 0, week 6 and week 13
Change in the Numerical Rating Scale (NRS) | Week 0, week 6 and week 13
Change in the Quality of life in late-stage dementia (QUALID) scale | Week -1, week 0, week 6 and week 13
Change in the EuroQoL Quality of Life Scale (EQ-5D) | Week -1, week 0, week 6 and week 13
Adverse events (AE) and serious adverse event (SAE) | Weeks 0-13
  Any AE or SAE will be recorded and treated as clinically appropriate throughout the study period.

OTHER OUTCOMES:
Change in the burden to personnel as measured by NPI-NH subscale | Week 0, week 6 and week 13

CONTACTS AND LOCATIONS:
Overall Officials: Bettina S Husebø, PhD, MD, Study Director — University of Bergen; Elisabeth Flo, PhD, Principal Investigator — University of Bergen; Ane Erdal, PhD candidate, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- [Derived] Erdal A, Flo E, Aarsland D, Ballard C, Slettebo DD, Husebo BS. Efficacy and Safety of Analgesic Treatment for Depression in People with Advanced Dementia: Randomised, Multicentre, Double-Blind, Placebo-Controlled Trial (DEP.PAIN.DEM). Drugs Aging. 2018 Jun;35(6):545-558. doi: 10.1007/s40266-018-0546-2. PMID 29725986
- [Derived] Blytt KM, Husebo B, Flo E, Bjorvatn B. Long-Term Pain Treatment Did Not Improve Sleep in Nursing Home Patients with Comorbid Dementia and Depression: A 13-Week Randomized Placebo-Controlled Trial. Front Psychol. 2018 Feb 13;9:134. doi: 10.3389/fpsyg.2018.00134. eCollection 2018. PMID 29487556